CLINICAL TRIAL: NCT03039374
Title: The Use of External Phase Array MRI, 3D Endoanal Ultrasound, and Manometry in the Diagnosis of Obstetric Anal Sphincter Injuries
Brief Title: External Phase MRI in Diagnosis of OASI
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Jaan Kirss, Principal Investigator, University of Turku
Other Study IDs: ISR-2014-10458
Record Dates: First submitted 2016-11-30; First posted 2017-02-01 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Anal Sphincter Injury; Obstetrics Trauma
Keywords: OASI; Faecal incontinence; Obstetric anal sphincter injury; MRI
MeSH Terms: conditions — Encopresis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OASI patients: All patients older than 18 and a 3rd or 4th degree perineal tear during birth meet the inclusion criteria. All women who have obtained such a injury during birth in the Vaasa or Seinäjoki Central hospitals will be evaluated for eligibility.
  Interventions: Other: Magnetic resonance imaging

INTERVENTIONS:
Other: Magnetic resonance imaging — The extent of obstetric anal sphincter injury will be evaluated using MRI, endoanal ultrasound and anal manometry

SUMMARY:
There is around 60 000 births annually in Finland. Around 1-5% of all vaginal deliveries in Finland complicate in a Grade III- IV perineal tear. Because the diagnosis of a sphincter lesion after birth can be challenging the total amount of women having obtained a sphincter lesion could be even grater.

The aim of our study is to compare different tools in the diagnosis of obstetric anal sphincter injury. In doing so the investigators hope to achieve early diagnosis of this pathology and thus facilitate early treatment of a possible sphincter defect.

DETAILED DESCRIPTION:
See the attacher research plan for a more detailed description

ELIGIBILITY:
Inclusion Criteria:

Women with OASI

Exclusion Criteria:

Under 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients older than 18 and a 3rd or 4th degree perineal tear observed during birth meet the inclusion criteria. All women who have obtained such a injury during birth in the Vaasa or Seinäjoki Central hospitals will be evaluated for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-09; Primary Completion 2017-09-20 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Comparison of MRI and endoanal ultrasound in diagnosis of obstetric anal sphincter injury | 6 months to 1 year
  Comparison of anal sphincter characteristics (length, thickness at 3 and 9 o'clock) and placement of the possible rupture with both imaging modalities

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Victorzon, prof., Study Director — Professor of surgery Turku University; Jaan Kirss, MD, Principal Investigator — Resident in Gastroenterological surgery

IPD SHARING:
Plan to Share IPD: No